CLINICAL TRIAL: NCT02364102
Title: Effect of Restoration of Euthyroidism in Patients With Primary Hypothyroidism on Brown Adipose Tissue Thermogenesis - the ThyroBAT Study
Brief Title: Effect of Hypothyroidism on Brown Adipose Tissue
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2015-028
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to study whether hypothyroidism negatively affects Brown adipose tissue (BAT) function in humans and whether BAT function can be restored to normal by thyroid hormone supplementation.

DETAILED DESCRIPTION:
Hypothyroidism is a frequent endocrine disorder, the prevalence of subclinical disease being 4.3% and of overt disease being 0.3%. Patients suffering from hypothyroidism frequently complain of increased cold sensitivity and involuntary weight gain, indicating changes in energy expenditure and response to cold challenge.

Recently, brown adipose tissue (BAT) has regained attention as an energy expending tissue. While it was previously thought to be of no or negligible relevance in human adults, recent studies clearly demonstrated the presence and metabolic activity of BAT in human adults. Upon activation of BAT by the sympathetic nervous system intracellular lipid stores are rapidly depleted. The generated free fatty acids fuel beta-oxidation and the respiratory chain within the mitochondria and activate at the same time uncoupling protein 1 (UCP1). This protein acts as a protonophore, allowing the flux of protons along the electrochemical gradient into the inner mitochondrial matrix instead of transferring their energy to adenosine triphosphate (ATP)-synthase. The short circuiting of the oxidative phosphorylation within the mitochondria leads to highly active cellular respiration and generation of heat. Basic research highlights the importance of thyroid hormone in the development and function of BAT.

It has recently been shown that hyperthyroidism exerts activating effects on BAT in adult humans.

The investigators aim to study whether hypothyroidism negatively affects BAT function in humans and whether BAT function can be restored to normal by thyroid hormone supplementation.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Serum thyroid-stimulating hormone (TSH) > 4.5 milli-International unit (mIU)/l
* body mass index (weight/height(m)²) 17.5 to 30 kg/m²

Exclusion Criteria:

* known concomitant disease influencing thyroid hormone metabolism
* chronic heart failure
* liver cirrhosis
* severe kidney failure
* metastasized cancer, except for thyroid cancer
* known hypersensitivity to cold, e.g. primary or secondary Raynaud's syndrome
* abuse of alcohol or illicit drugs
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: currently hypothyroid patients which are started on levothyroxin substitution
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
difference in cold induced thermogenesis between baseline and restoration of euthyroidism, assessed as the increase in resting energy expenditure after a mild cold stimulus determined by indirect calorimetry | before and after 3 months after restoration of euthyroidism

SECONDARY OUTCOMES:
difference in supraclavicular skin temperature (before and after cold exposure) | before and after 3 months after restoration of euthyroidism
levels of Irisin in serum | before and after 3 months after restoration of euthyroidism
patient's perception of cold | before and after 3 months after restoration of euthyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, Principal Investigator — Department of Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided